CLINICAL TRIAL: NCT07395596
Title: A Prospective, Randomized Controlled Clinical Study of the Effect of Remimazolam on the Incidence of Hypoxia in High-risk Patients Undergoing Painless Tracheoscopy
Brief Title: Remimazolam for Bronchoscopy in High-Risk Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shaoxing People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Yueying Zheng, Vice Director of the Department of Anesthesiology, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZJU2026B0127
Record Dates: First submitted 2025-07-07; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Infection; Pulmonary Nodule; Phthisis; Endotracheal Tumour; Lymphadenectasis
Keywords: hypoxia; remimazolam; propofol; fiberoptic bronchoscopy
MeSH Terms: conditions — Tuberculosis, Pulmonary; Hypoxia | interventions — Propofol; Alfentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The propofol - alfentanil group（The control group） (Active Comparator): In this group, general anesthesia was administered using the classic propofol and alfentanil. The patients underwent fiberoptic bronchoscopy while maintaining spontaneous breathing and with a MOAA/S score of ≤2.
  Interventions: Drug: propofol and alfentanil
- The remimazolam and propofol - alfentanil group (The experimental group) (Experimental): This group received general anesthesia with remimazolam combined with propofol for sedation and alfentanil. Fiberoptic bronchoscopy was done while patients maintained spontaneous breathing and had a MOAA/S score of ≤2.
  Interventions: Drug: remimazolam combined with propofol and alfentanil

INTERVENTIONS:
Drug: propofol and alfentanil — General anesthesia with spontaneous breathing maintained is administered using propofol and alfentanil.
  Arms: The propofol - alfentanil group（The control group）
Drug: remimazolam combined with propofol and alfentanil — General anesthesia with spontaneous breathing maintained is administered using remimazolam combined with propofol and alfentanil.
  Arms: The remimazolam and propofol - alfentanil group (The experimental group)

SUMMARY:
Bronchoscopy is currently widely used for the diagnosis and treatment of various respiratory diseases. However, the operation of bronchoscopy is irritating, causes a strong stress response, and shares the airway with the patient, making the patient highly susceptible to respiratory and cardiovascular risks. Among these risks, hypoxia is the most common adverse event.Different drug regimens can be selected for anesthesia under deep sedation. The combination of analgesic agents can help reduce coughing during bronchoscopy. Therefore, we employ a combination of sedative and analgesic drugs for painless bronchoscopy procedures. Among sedatives, propofol is the most commonly used. However, due to its disadvantages, such as respiratory and circulatory depression, we have introduced a novel approach combining remimazolam for sedation. The aim is to investigate whether this new regimen, compared to traditional propofol-based sedation, can reduce the incidence of hypoxia, minimize circulatory depression, and lead to faster postoperative awakening and recovery. Additionally, we hope to observe fewer adverse events, such as perioperative nausea and vomiting, excessive secretions, dizziness, and chills.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class Ⅲ - Ⅳ
* Scheduled for elective painless bronchoscopy -

Exclusion Criteria:

* Age < 18 years
* Patients who are uncooperative（e.g. due to mental illness）
* Patients who are on chronic use of opioids, benzodiazepine - class hypnotics, or antidepressants
* Patients with a history of allergy to the anesthetics used
* Patients who are anticipated to have a difficult airway
* Body mass index（BMI）<18.5kg/m² or >30kg/m²
* Preoperative oxygen saturation <92% while breathing room air
* Other：Patients who are deemed by the investigator to be unsuitable for participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia（75% ≤ SpO2 < 90% for <60 s） | Periprocedural

SECONDARY OUTCOMES:
The incidence of severe hypoxia（SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s） | Periprocedural
Non-Invasive Blood Pressure changes: The area under the curve (AUC) of the patient's mean blood pressure over time from pre-anesthesia induction to the end of bronchoscopy during patient monitoring | Periprocedural
The area under the curve (AUC) of the patient's mean blood pressure during observation in Post-Anesthesia Care Unit | Periprocedural
The dosage of vasoactive drugs administered. | Periprocedural

OTHER OUTCOMES:
The incidence of other adverse events | Periprocedural
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affliated Hospital, Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Shaoxing City First People's Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol